CLINICAL TRIAL: NCT00420966
Title: Phase IV Study of Respiratory Syncytial Virus Monoclonal Antibody Therapy in High-risk Infants and Toddlers
Brief Title: Utilization and Compliance of Respiratory Syncytial Virus Monoclonal Antibody Therapy
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 456-2005
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2017-09

CONDITIONS: Lower Respiratory Tract Infection; Respiratory Syncytial Virus Infections
Keywords: lower respiratory tract infection; respiratory syncytial virus infections; palivizumab; outcomes; utilization; compliance
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Patient Acceptance of Health Care; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the utilization patterns and compliance rates of palivizumab, which is a monoclonal antibody therapy used to prevent respiratory syncytial virus infection.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is the most important viral respiratory pathogen in children. Infection due to RSV represents a large public health burden; in Canada, it accounts for 5,800 hospitalizations annually. The peak incidence of RSV disease occurs between 2-6 months of age with half of all infants infected in the first year of life. Palivizumab has been approved for the prevention of serious lower respiratory tract disease caused by RSV in pediatric patients at high-risk of RSV disease. These children include those born premature, those with bronchopulmonary dysplasia (BPD), and those with hemodynamically significant congenital heart disease (CHD).

With the recent approval of palivizumab in Canada, access to this medication has increased. However, there are limited data on utilization, compliance, and health outcomes, particularly the frequency and severity of RSV infections. The primary objective of this study is to provide insight into the current management (utilization, compliance) of children at high-risk of RSV infection with palivizumab prophylaxis in the tertiary care centers and community settings through the development of a Canadian Registry Database.

ELIGIBILITY:
Inclusion Criteria:

* All children who receive at least one dose of palivizumab

Exclusion Criteria:

* The child's parent or legal guardian could not communicate in either English or French
* The child had received palivizumab as part of a clinical trial during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children who have received at least one dose of palivizumab.
Sampling Method: Non-Probability Sample
Enrollment: 25003 (Actual)
Dates: Start 2005-10; Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Determine palivizumab outcome measures | Per respiratory syncytial virus season
  The objectives of this study are:
  * To determine palivizumab usage patterns, annually
  * To understand palivizumab infant demographics, including: potential neonatal, familial and environmental risk factors
  * To determine reasons for hospitalization, respiratory syncytial virus hospitalization rates, length of stay, morbidity and mortality
  * To determine intensive care unit admissions, length of stay, use of respiratory support (e.g., mechanical ventilation, CPAP) and complication rates
  * To determine compliance rates
  * To collect safety data

CONTACTS AND LOCATIONS:
Overall Officials: Ian Mitchell, MB, FRCPC, Principal Investigator — University of Calgary; Krista L Lanctôt, PhD, Study Director — Sunnybrook Health Sciences Centre; Bosco Paes, MD, FRCPC, Study Director — McMaster University
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - McMaster Children's Hospital, Hamilton, Ontario

REFERENCES:
- [Result] Mitchell I, Paes BA, Li A, Lanctot KL; CARESS investigators. CARESS: the Canadian registry of palivizumab. Pediatr Infect Dis J. 2011 Aug;30(8):651-5. doi: 10.1097/INF.0b013e31821146f7. PMID 21343842
- [Result] Paes B, Mitchell I, Li A, Lanctot KL; CARESS Investigators. A comparative study of respiratory syncytial virus (RSV) prophylaxis in premature infants within the Canadian Registry of Palivizumab (CARESS). Eur J Clin Microbiol Infect Dis. 2012 Oct;31(10):2703-11. doi: 10.1007/s10096-012-1617-7. Epub 2012 May 1. PMID 22546928
- [Result] Paes B, Mitchell I, Yi H, Li A, Lanctot KL; CARESS Investigators. Hospitalization for respiratory syncytial virus illness in Down syndrome following prophylaxis with palivizumab. Pediatr Infect Dis J. 2014 Feb;33(2):e29-33. doi: 10.1097/INF.0000000000000019. PMID 23989104
- [Result] Yi H, Lanctot KL, Bont L, Bloemers BL, Weijerman M, Broers C, Li A, Kiss A, Mitchell I, Paes B; CARESS investigators. Respiratory syncytial virus prophylaxis in Down syndrome: a prospective cohort study. Pediatrics. 2014 Jun;133(6):1031-7. doi: 10.1542/peds.2013-3916. Epub 2014 May 5. PMID 24799541
- [Result] Chen JJ, Chan P, Paes B, Mitchell I, Li A, Lanctot KL; CARESS investigators. Serious Adverse Events in the Canadian Registry of Children Receiving Palivizumab (CARESS) for Respiratory Syncytial Virus Prevention. PLoS One. 2015 Aug 3;10(8):e0134711. doi: 10.1371/journal.pone.0134711. eCollection 2015. PMID 26237402
- [Result] Chan P, Li A, Paes B, Abraha H, Mitchell I, Lanctot KL; CARESS investigators. Adherence to Palivizumab for Respiratory Syncytial Virus Prevention in the Canadian Registry of Palivizumab. Pediatr Infect Dis J. 2015 Dec;34(12):e290-7. doi: 10.1097/INF.0000000000000922. PMID 26780032
- [Result] Hui C, Paes B, Papenburg J, Mitchell I, Li A, Lanctot KL; CARESS Investigators. Palivizumab Adherence and Outcomes in Canadian Aboriginal Children. Pediatr Infect Dis J. 2016 Nov;35(11):1187-1193. doi: 10.1097/INF.0000000000001282. PMID 27331856
- [Result] Paes B, Mitchell I, Li A, Harimoto T, Lanctot KL. Respiratory-related hospitalizations following prophylaxis in the Canadian registry for palivizumab (2005-2012) compared to other international registries. Clin Dev Immunol. 2013;2013:917068. doi: 10.1155/2013/917068. Epub 2013 Jun 19. PMID 23861694
- [Result] Paes B, Mitchell I, Li A, Lanctot KL. Respiratory hospitalizations and respiratory syncytial virus prophylaxis in special populations. Eur J Pediatr. 2012 May;171(5):833-41. doi: 10.1007/s00431-011-1654-8. Epub 2011 Dec 28. PMID 22203430
- [Result] Manzoni P, Paes B, Lanctot KL, Dall'Agnola A, Mitchell I, Calabrese S, Maule M, Girardi E, Harimoto T, Li A. Outcomes of Infants Receiving Palivizumab Prophylaxis for Respiratory Syncytial Virus in Canada and Italy: An International, Prospective Cohort Study. Pediatr Infect Dis J. 2017 Jan;36(1):2-8. doi: 10.1097/INF.0000000000001340. PMID 27649365
- [Result] Wang DY, Li A, Paes B, Mitchell I, Lanctot KL; CARESS Investigators. First versus second year respiratory syncytial virus prophylaxis in chronic lung disease (2005-2015). Eur J Pediatr. 2017 Mar;176(3):413-422. doi: 10.1007/s00431-017-2849-4. Epub 2017 Jan 20. PMID 28105526
- [Result] Li A, Wang DY, Lanctot KL, Mitchell I, Paes BA; CARESS Investigators. Comparing First- and Second-year Palivizumab Prophylaxis in Patients With Hemodynamically Significant Congenital Heart Disease in the CARESS Database (2005-2015). Pediatr Infect Dis J. 2017 May;36(5):445-450. doi: 10.1097/INF.0000000000001357. PMID 28403044
- [Result] Bjornson C, Chan P, Li A, Paes B, Lanctot KL, Mitchell I. Palivizumab prophylaxis for respiratory syncytial virus in infants with cystic fibrosis: is there a need? Eur J Clin Microbiol Infect Dis. 2018 Jun;37(6):1113-1118. doi: 10.1007/s10096-018-3225-7. Epub 2018 Mar 19. PMID 29557081
- [Derived] Paes BA, Saleem M, Li A, Lanctot KL, Mitchell I; CARESS Investigators. Respiratory Syncytial Virus Prophylaxis in Immunocompromised Children: Outcomes From the Canadian RSV Evaluation Study of Palivizumab Registry Over Twelve Seasons (2005-2017). Pediatr Infect Dis J. 2020 Jun;39(6):539-545. doi: 10.1097/INF.0000000000002665. PMID 32235248
- [Derived] Paes B, Li A, Kim D, Lanctot KL, Mitchell I; CARESS Investigators. A Comparison of Respiratory Syncytial Viral Prophylaxis in Multiple Births versus Singletons in the Canadian Registry of Palivizumab. Am J Perinatol. 2021 Aug;38(S 01):e129-e136. doi: 10.1055/s-0040-1708804. Epub 2020 Mar 31. PMID 32232817
- [Derived] Wang DY, Saleem M, Paes BA, Mitchell I, Li A, Lanctot KL; CARESS Investigators. Respiratory Syncytial Virus Prophylaxis in Neurologic and Muscular Disorders in the Canadian Respiratory Syncytial Virus Evaluation Study of Palivizumab. Pediatr Infect Dis J. 2019 Aug;38(8):775-780. doi: 10.1097/INF.0000000000002297. PMID 30985509
- [Derived] Kim D, Saleem M, Paes B, Mitchell I, Lanctot KL. Respiratory Syncytial Virus Prophylaxis in Infants With Congenital Diaphragmatic Hernia in the Canadian Respiratory Syncytial Virus Evaluation Study of Palivizumab, 2005-2017. Clin Infect Dis. 2019 Aug 30;69(6):980-986. doi: 10.1093/cid/ciy1010. PMID 30517603